CLINICAL TRIAL: NCT05779943
Title: Strategy to Reduce Bladder Activity With RhPSMA 7.3: Comparison of 18F-RhPSMA 7.3 PET/CT With and Without Furosemide in Biochemical Recurrence of Prostate Cancer
Brief Title: Comparison of 18F-rhPSMA-7.3 PET/CT With and Without Furosemide in Biochemical Recurrence of Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Blue Earth Diagnostics (Industry)
Responsible Party: Principal Investigator, David M Schuster, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00004720; RAD5689-22-BED-IIT-439 (Other: Emory University Hospital/Winship Cancer Institute); STUDY00004720 (Other: Emory University Hospital/Winship Cancer Institute); NCI-2023-01322 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA138292 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-03-22 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Furosemide; Magnetic Resonance Spectroscopy; X-Rays; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT) (Experimental): Patients receive F-18 rhPSMA 7.3 tracer IV and then undergo PET-CT scans with and without furosemide IV on study.
  Interventions: Drug: Furosemide; Other: F18-rhPSMA-7.3; Procedure: Positron Emission Tomography; Procedure: Computed Tomography

INTERVENTIONS:
Drug: Furosemide — Given IV
  Other Names: 54-31-9, FRS, Furosemide, FUROSEMIDE, Lasix, Lasix, LB 502, LB-502, LB-502, SK-Furosemide
Other: F18-rhPSMA-7.3 — Given IV
  Other Names: (18F)-rhPSMA-7.3,18F-rhPSMA-7.3,18FrhPSMA-7.3,2305081-64-3,F-18-rhPSMA-7.3,FLOTUFOLASTAT F-18, Fluorine F18 radiohybrid PSMA-7.3, Fluorine F18 rhPSMA-7.3, Fluorine-18 rhPSMA-7.3, rhPSMA-7.3(18F)
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging,Positron Emission Tomography, PET, PET SCAN
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT, CAT Scan, CAT scan, CAT Scan,Computed Axial Tomography,Computed Tomography, Computerized Axial Tomography

SUMMARY:
This phase II trial evaluates Fluorine-18 radiohybrid prostate-specific membrane antigen (18F- rhPSMA)-7.3 positron emission tomography (PET)/computed tomography (CT) scans with and without furosemide for the reduction of bladder activity in patients with prostate cancer that has come back (recurrent) based on elevated levels of prostate-specific antigen (PSA) in the blood (biochemical) after prostate surgery (prostatectomy). Furosemide is a diuretic substance that increases the urine flow into the bladder, thereby decreasing the level of radioactivity within the bladder, which may help to see any abnormal areas that could be masked by the radioactivity within the bladder. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, rhPSMA ligand. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. Adding furosemide to 18F-rhPSMA 7.3 PET/CT scans may help to better detect and treat patients with biochemically recurrent prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if administering 20 mg furosemide intravenously (IV) at the time of radiotracer injection significantly reduces bladder activity compared with the same patient scanned without furosemide as internal control.

SECONDARY OBJECTIVES:

I. To compare detection rates of recurrent disease in blinded interpretations between the furosemide and non-furosemide 18FrhPSMA-7.3 PET/CT scans, with patients serving as their own internal controls.

II. To compare reader confidence in identifying prostate bed and other recurrent lesions on a 18F-rhPSMA-7.3 PET/CT with furosemide compared with 18F-rhPSMA-7.3 PET/CT without furosemide.

OUTLINE:

Patients receive 18F-rhPSMA 7.3 tracer IV and then undergo PET-CT scans with and without furosemide IV on study.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate, post-prostatectomy
* Biochemical recurrence of prostate cancer following radical prostatectomy (RP) with or without adjuvant or salvage therapy: PSA >= 0.2 ng/mL followed by a subsequent confirmatory PSA value >= 0.2 ng/mL
* Age over 18
* Ability to provide written informed consent
* Patients with standard of care creatinine =< 1.3 mg/dL performed within 90 days prior to enrollment

Exclusion Criteria:

- Inability to undergo 18F-rhPSMA PET-CT, contraindications to furosemide or urinary incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2028-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charles V. Marcus, MBBS, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide followed by without furosemide .: Patients receive F-18 rhPSMA 7.3 tracer IV and then undergo PET-CT scans with and without furosemide IV on study.
  Furosemide: Given IV
  F18-rhPSMA-7.3: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
  Computed Tomography: Undergo PET/CT scan
- Group B - Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide followed by with furosemide.: Patients receive F-18 rhPSMA 7.3 tracer IV and then undergo PET-CT scans without and with furosemide IV on study.
  Furosemide: Given IV
  F18-rhPSMA-7.3: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
  Computed Tomography: Undergo PET/CT scan
Period: V1 (1-30 days after consent/screening)
Arm/Group | Group A - Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide followed by without furosemide . | Group B - Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide followed by with furosemide.
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: V2 (2-7days after PET/CT #1)
Arm/Group | Group A - Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide followed by without furosemide . | Group B - Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide followed by with furosemide.
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.95 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Bladder Activity as Measured by Bladder Standardized Uptake Value (SUV) Mean
Description: Change in bladder SUV mean will be assessed using a paired t-test, or using a non-parametric equivalent such as a Wilcoxon signed rank test. Descriptively, change in bladder SUV mean will be reported for those administered 20 mg furosemide intravenously (IV) at the time of radiotracer injection first (group A), and those administered 20mg furosemide IV at the time of radiotracer injection second (group B).
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- Without furosemide: Patients receive F-18 rhPSMA 7.3 tracer IV and then undergo PET-CT scans with and without furosemide IV on study.
  Furosemide: Given IV
  F18-rhPSMA-7.3: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
  Computed Tomography: Undergo PET/CT scan
Arm/Group | Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT) | Without furosemide
Number analyzed (Participants) | 20 | 20
SUV | 3.9 (3.71) | 20.64 (31.50)

2. Secondary Outcome: Change in Bladder and Renal Activity (Kidney SUV)
Description: Kidney SUV - Change in bladder and renal activity will be assessed using paired t-tests, or using non-parametric equivalents such as a Wilcoxon signed rank tests. Descriptively, bladder and renal activity will be reported for those administered 20 mg furosemide IV at the time of radiotracer injection first (group A), and those administered 20 mg furosemide IV at the time of radiotracer injection second (group B).
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT) | Without furosemide
Number analyzed (Participants) | 20 | 20
SUV | 24.87 (7.95) | 27.12 (8.46)

3. Secondary Outcome: Change in Bladder and Renal Activity (Bladder Volume, ML)
Description: (Bladder Volume, ML) - Change in bladder and renal activity will be assessed using paired t-tests, or using non-parametric equivalents such as a Wilcoxon signed rank tests. Descriptively, bladder and renal activity will be reported for those administered 20 mg furosemide IV at the time of radiotracer injection first (group A), and those administered 20 mg furosemide IV at the time of radiotracer injection second (group B).
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: ML
Arm/Group | Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT) | Without furosemide
Number analyzed (Participants) | 20 | 20
ML | 300.22 (151.30) | 147.69 (172.31)

4. Secondary Outcome: Recurrent Disease Rate
Description: Defined as presence of unequivocal soft tissue radiotracer uptake that is characteristic of malignancy in the prostate bed and/or surrounding soft tissues and within pelvic lymph nodes. Recurrent disease rates will be compared (furosemide versus non-furosemide flotufolastat F-18 radiohybrid prostate-specific membrane antigen (18F-rhPSMA)-7.3 positron emission tomography (PET) scans using McNemar's tests. Rates will be reported, along with 95% exact confidence intervals using the Clopper-Pearson method. Descriptively, recurrent disease rate will be reported for those administered 20 mg furosemide IV at the time of radiotracer injection first (group A), and those administered 20 mg furosemide IV at the time of radiotracer injection second (group B).
Time Frame: Up to 2 weeks
Measure: Number; unit: Participants
Arm/Group | Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT) | Without furosemide
Number analyzed (Participants) | 20 | 20
Participants
  Prostate bed - Negative (No recurrence detected) | 3 | 8
  Prostate bed - Positive (Recurrence detected) | 17 | 12
  Pelvic - Negative (No recurrence detected) | 18 | 17
  Pelvic - Positive (Recurrence detected) | 2 | 3
  Extra pelvic - Negative (No recurrence detected) | 16 | 16
  Extra pelvic - Positive (Recurrence detected) | 4 | 4
  Patient level - Negative (No recurrence detected) | 2 | 5
  Patient level - Positive (Recurrence detected) | 18 | 15

5. Secondary Outcome: Reader Confidence Score
Description: The readers' confidence in identifying prostate bed, pelvic and retroperitoneal nodal disease and other recurrence on 18F-rhPSMA-7.3 PET/computed tomography (CT) with furosemide compared with the 18F-rhPSMA-7.3 PET/CT without furosemide will be scored using a 5-point Likert scale ( 1 - Definitely benign, 2- probably benign, 3 - equivocal, 4 - probably malignant, 5 - definitely malignant). This analysis will be descriptive, with summary statistics reported with and without furosemide. Variables will be summarized using frequencies and percentages. In our analysis, 1,2 (no) will be considered benign while 3,4,5 malignant (yes). A high Likert score indicates that the reader is confident that the finding on the imaging is cancer (worse outcome), while a low score indicates no cancer (better outcome). All tests will be two-sided with an alpha level of 0.05, unless otherwise noted. Statistical analysis will be conducted using SAS 9.4.
Time Frame: 1 Month
Measure: Number; unit: participants
Arm/Group | Treatment (furosemide, F-18 rhPSMA-7.3, PET-CT) | Without furosemide
Number analyzed (Participants) | 20 | 20
participants
  Prostate Agree (Yes) (High Lickert Score 3-5) | 10 | 9
  Prostate Agree (No) (Low Lickert Score 1-2) | 10 | 11
  Pelvis-Agree (Yes) (High Lickert Score 3-5) | 19 | 19
  Pelvis-Agree (No) (Low Lickert Score 1-2) | 1 | 1
  Extra-Prostate-Agree (Yes) (High Lickert Score 3-5) | 15 | 15
  Extra-Prostate-Agree (No) (Low Lickert Score 1-2) | 5 | 5

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide Study Visit 1 (1-30 days after consent/screening); Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide Study Visit 2 (2-7days after PET/CT #1): Patients receive F-18 rhPSMA 7.3 tracer IV and then undergo PET-CT scans with furosemide IV on study.
  Furosemide: Given IV
  F18-rhPSMA-7.3: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
  Computed Tomography: Undergo PET/CT scan
- Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide Study Visit 2 (2-7days after PET/CT #1); Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide Visit 1 (1-30 days after consent/screening): Patients receive F-18 rhPSMA 7.3 tracer IV and then undergo PET-CT scans without furosemide IV on study.
  Furosemide: Given IV
  F18-rhPSMA-7.3: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
  Computed Tomography: Undergo PET/CT scan
Arm/Group | Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide Study Visit 1 (1-30 days after consent/screening) | Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide Study Visit 2 (2-7days after PET/CT #1) | Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide Visit 1 (1-30 days after consent/screening) | Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide Study Visit 2 (2-7days after PET/CT #1)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide Study Visit 1 (1-30 days after consent/screening) (N=10) | Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide Study Visit 2 (2-7days after PET/CT #1) (N=10) | Complete 18F-rhPSMA-7.3 PET/CT #1 without furosemide Visit 1 (1-30 days after consent/screening) (N=10) | Complete 18F-rhPSMA-7.3 PET/CT #1 with furosemide Study Visit 2 (2-7days after PET/CT #1) (N=10)
Bruising at injection site (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT05779943/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT05779943/ICF_001.pdf